CLINICAL TRIAL: NCT01740622
Title: Healthy Homes Healthy Children (H3C)
Acronym: H3C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012-2903
Record Dates: First submitted 2012-10-19; First posted 2012-12-04 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Injury in the Home
Keywords: Injury; Injury Prevention; Cincinnati Home Injury Prevention; Injury Hazards; Modifiable Injury Hazards
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Injury Intervention Group (Experimental): In homes of children who are randomized to the injury intervention arm of the trial, a comprehensive survey of injury hazards in living spaces will be undertaken. In addition to quantifying hazards, the area of living spaces will be obtained to allow the determination of both the number and density (number of hazards per 100 sq.ft.) of injury hazards. If one or more injury hazards are identified, they will be removed and/or modified to reduce exposure and injury risk. The intervention is focused on areas in living spaces below 1-meter (~39 inches) in height from (the 75th percentile in height or eye-level for a 3-year old US male toddler) which might be easily reached or climbed on by children less than 4 years.
  Interventions: Other: Injury Prevention Measures
- Control Group (No Intervention): Participants who are assigned to the control group will have their medical claims examined related to injury in the home. Households in this control condition will also be provided with information sheets on child safety developed by the American Academy of Pediatrics, The Injury Prevention Program (TIPP). These age-based recommendations for child safety are provided as standard of care at many pediatric offices.

INTERVENTIONS:
Other: Injury Prevention Measures — The hazards identified in the home will be reviewed with the parent and the proposed interventions will be presented. Intervention options are designed and prioritized so that the most passive and durable interventions are recommended first (e.g. self-closing, self-locking stair gate) and progressively less 'passive' and less durable options last (e.g. area gate, pressure mounted gate, or refusal of intervention).
  Other Names: Injury in the Home; Injury; Injury Prevention; Cincinnati Home Injury Prevention; Injury Hazards; Modifiable Injury Hazards
  Arms: Injury Intervention Group

SUMMARY:
Aim

To evaluate the efficacy of a CCHMC Human Resources Benefits program to reduce exposure to injury hazards and subsequent injury-related medical claims for their children.

Hypothesis

H1: The investigators anticipate, based on our recently completed trial, that the installation of multiple, passive safety devices in the homes of children 6- to 36-month old children of CCHMC non-contract employees randomized to the intervention group will reduce childhood injuries and medical claims by 50% compared to children of CCHMC non-contract employees who do not receive the home safety program.

H2: Cincinnati Children's Hospital Medical Center Employees whose children are randomized to the intervention will have 30% less lost work days compared to employees whose children are assigned control group.

DETAILED DESCRIPTION:
Injury is the leading cause of morbidity and mortality for US children; the home is the leading location of injury for younger US children. Unintentional injuries in the home environment account for more than 4 million visits to emergency departments, with over 74,000 hospitalizations and 2,800 deaths each year in US children at a cost in excess of $3 billion annually and $800 per emergency visit. Ambulatory visit rates for injury in US Children are more than 3-fold higher than emergency visit rates and account for more than 13 million visits to offices and clinics each year in the U.S.

There is increasing interest in developing systems to improve the health of populations of children residing in the Cincinnati Children's Hospital Medical Center (CCHMC) primary service area. Emerging payment models are fostering programs that can improve proactive population health management including preventive measures to reduce morbidity and improve the value of health services provided by insurers and accountable care organizations. This project will test the efficacy of an intervention to reduce exposure to injury hazards in the home and subsequent preventable and medically attended injury in young children.

Experimental Group: In homes of children randomized to the intervention arm of the trial, a comprehensive observational survey of living spaces will be undertaken. The study will examine living spaces to which a child may be exposed including 5 high-exposure, high-risk areas (main activity room, kitchen, child's bedroom and bathrooms, and stairways). In addition to quantifying hazards, the area of rooms will be obtained allowing for determination of both the number and density of injury hazards.

The hazards identified by the intervention team will be reviewed with the parent and the proposed interventions will be presented. Intervention options are designed and prioritized so that the most passive and durable interventions are recommended first and progressively less 'passive' and less durable options last. After consent is obtained, passive measures will be installed across the living space as indicated.

Control Group: Participants who are assigned to the control group will have their medical claims examined related to injury in the home. Households in this control condition will also be provided with information sheets on child safety developed by the American Academy of Pediatrics, The Injury Prevention Program (TIPP). These age-based recommendations for child safety are provided as standard of care at many pediatric offices.

ELIGIBILITY:
Inclusion Criteria:

* Current CCHMC qualified beneficiaries (non-contract workers)
* Child is both covered by a CCHMC health insurance plan and is less than 8 months of age at the time of screening
* Employees must be at least 18 years of age
* Employee must have no plans to leave CCHMC employment within next 12 months
* Employee must have no plans to relocate greater than 90 minutes away from CCHMC in the next 12 months
* Employees must speak fluent English

Exclusion Criteria:

* The child is greater than 8 months of age at time of screening
* Employee is non-English speaking
* Not a current CCHMC employee
* Child not covered by CCHMC health insurance plan
* Employees who are not 18 years of age
* Live beyond a 90-minute driving radius from Cincinnati Children's Hospital or have plans to relocate outside of a 90-minute driving radius from Cincinnati Children's Hospital in the next 12 months at the time of screening
* Have plans to leave employment at Cincinnati Children's Hospital in the next 12 months at the time of screening

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 520 (Actual)
Dates: Start 2012-10; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Any modifiable and medically-attended injury in enrolled children sustained in the home | Quarterly ( quarterly online surveys) (up to 24 months)
  The primary outcome measure will be claims for medically-attended injury sustained in the home environment. This composite outcome includes any medical claims from phone calls, office, clinic, and emergency department (ED) visits by enrolled children in the home for injuries whose exposure was modified by the installed safety devices (i.e. falls, cuts/pierces, struck/strike, burns, poisonings).

SECONDARY OUTCOMES:
Presenteeism / Absenteeism at work due to child's injury | Quarterly (online surveys) (up to 2 years)
  Furthermore, the investigators will attempt to capture work loss, presenteeism and absenteeism associated with medical treatment for a child's injury.

CONTACTS AND LOCATIONS:
Overall Officials: Kiernan Phelan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States